CLINICAL TRIAL: NCT02679898
Title: The Effect of the Combination of Whole Body Vibration and External Load Exercise Training on Cardiovascular and Autonomic Function in Obese Individuals
Brief Title: Whole Body Vibration and External Load Exercise Training on Cardiovascular and Autonomic Function in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HSC201311173
Record Dates: First submitted 2016-02-01; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: Arterial function; Whole-body vibration training; Aortic blood pressures; Wave reflection; Muscle strength; Endothelial function; Blood flow
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lean Control (No Intervention): This arm involves not making any changes to the subject's lifestyle at the moment of the start of the intervention and for 6 weeks.
- Overweight/Obese Control (No Intervention): This arm involves not making any changes to the subject's lifestyle at the moment of the start of the intervention and for 6 weeks.
- Unloaded-Whole Body Vibration (WBVT) (Experimental): Lower-body exercise training on a vibration platform
  Interventions: Other: Unloaded-Whole Body Vibration (WBVT)
- Loaded-Whole Body Vibration (WBVT) (Experimental): Externally loaded lower-body exercise training on a vibration platform
  Interventions: Other: Loaded-Whole Body Vibration (WBVT)

INTERVENTIONS:
Other: Unloaded-Whole Body Vibration (WBVT) — The unloaded-WBVT intervention consists of four leg exercises performed dynamically over a vibrating platform 3 times/week for 6 weeks. Dynamic movements were performed with controlled movements starting from an upright position into a 90 and 120 degree knee angle, wide-stance squat, and maximal heel elevation. The training volume increased progressively by increasing the intensity of the vibration (30-35 Hz; low-high amplitude), duration of exercise (30-60 sec), number of sets per exercise (2-8), and total during of training session, while decreasing the rest periods (60-30 sec).
  Arms: Unloaded-Whole Body Vibration (WBVT)
Other: Loaded-Whole Body Vibration (WBVT) — The loaded-WBVT intervention consists of four leg exercises performed dynamically over a vibrating platform 3 times/week for 6 weeks. Importantly, an external load was applied to a weight vest to account for the necessary weight to perform a specific number of repetitions (progressed from 15-8 repetitions maximum during the 6 weeks). Dynamic movements were performed with controlled movements starting from an upright position into a 90 and 120 degree knee angle, wide-stance squat, and maximal heel elevation. The training volume increased progressively by increasing the intensity of the vibration (30-35 Hz; low-high amplitude), duration of exercise (30-60 sec), number of sets per exercise (2-8), and total during of training session, while decreasing the rest periods (60-30 sec).
  Arms: Loaded-Whole Body Vibration (WBVT)

SUMMARY:
Obesity is directly related to arterial dysfunction and negatively associated to muscle strength. High-intensity resistance exercise is the favored modality to offset muscle weakness, yet, adverse effects on arterial function (pulse wave velocity, wave reflection, and aortic and brachial blood pressures) have been observed. Conventional unloaded-whole body vibration training (WBVT) has improved arterial function in overweight/obese women but appears to be low-intensity. Nevertheless, the effects of moderate-intensity (by adding external load) WBVT on arterial and muscle function are unknown. Therefore, the purpose of this study was to examine whether loaded-WBVT would induce greater benefits than unloaded-WBVT on arterial and muscle function in young overweight/obese women. Furthermore, we examined whether these changes were similar to healthy lean young women.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effects of 6 weeks of loaded-WBVT on arterial stiffness, peripheral and aortic blood pressures, wave reflection, endothelial function, and muscle strength in overweight/obese women.

The specific aims of the study were:

1. To examine whether 6 weeks of loaded-WBVT was more beneficial than unloaded-WBVT in decreasing cardiovascular risk factors by assessing arterial stiffness (aortic, leg, and systemic), aortic blood pressures and wave reflection, brachial blood pressures, autonomic function, endothelial function, and blood flow (leg and arm).
2. To determine the extent to which 6 weeks of loaded-WBVT improved body composition measured by changes in fat and lean mass utilizing dual-energy x-ray absorptiometry and waist circumference.
3. To evaluate the effect of 6 wees of loaded-WBVT on muscle strength by using the one-repetition maximum test (leg press and chest press exercises).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 to 25 years of age
* Sedentary (less than 120 min per wk)
* 15 lean (Body mass index of 18-25 kg/m²)
* 45 overweight/obese (Body mass index of 27-39.9 kg/m²)

Exclusion Criteria:

* Younger than 18 or older than 25 years of age
* Body mass index lower than 18 or higher than 39.9
* Physically active or competitively active
* Smokers
* Pregnant
* Irregular menstrual cycle
* Use of dietary supplementations (e.g.,L-arginine,L-citrulline,antioxidants)
* Any contraindications to exercise and/or whole-body vibration exercise

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | 6 weeks
  Aortic, leg, and systemic pulse wave velocity acquired through non-invasive sensors.
Pressure Wave Reflection | 6 weeks
  Augmentation index acquired through radial tonometry.

SECONDARY OUTCOMES:
Body Composition | 6 weeks
  Measuring fat mass and lean mass from dual-energy x-ray absorptiometry.
Muscle Strength | 6 weeks
  Using one-repetition maximum (1-RM) test for the leg press and chest press exercises.
Autonomic Function | 6 weeks
  Heart rate variability through electrocardiogram.
Blood Pressures | 6 weeks
  Non-invasive measures of brachial and aortic blood pressures.
Endothelial Function | 6 weeks
  Non-invasive arm and leg blood flow using vascular ultrasound positioned on my skin at rest and during increased blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Principal Investigator — Florida State University
Locations (1):
- FSU College of Human Sciences, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez-Alvarado S, Jaime SJ, Ormsbee MJ, Campbell JC, Post J, Pacilio J, Figueroa A. Benefits of whole-body vibration training on arterial function and muscle strength in young overweight/obese women. Hypertens Res. 2017 May;40(5):487-492. doi: 10.1038/hr.2016.178. Epub 2017 Jan 12. PMID 28077859